CLINICAL TRIAL: NCT00524472
Title: The Effect of Hyperinsulinemic Glucose Control on Outcomes Following Cardiac Surgery
Brief Title: Outcomes Study of Hyperinsulinemic Glucose Control in Cardiac Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 07-470
Record Dates: First submitted 2007-08-31; First posted 2007-09-03 (Estimated); Results first posted 2018-10-26 (Actual); Last update posted 2018-10-26 (Actual); Status verified 2018-02

CONDITIONS: Cardiac Surgery
Keywords: Hyperinsulinemic glucose control; cardiac surgery; Outcome
MeSH Terms: interventions — Constriction; Insulin

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Hyperinsulinemic-normoglycemic clamp (Experimental): Patients will be randomized to receive the hyperinsulinemic-normoglycemic clamp titrating the blood glucose to 80-110 mg/dL.
  Interventions: Other: Hyperinsulinemic-normoglycemic clamp
- Insulin at the standard of care levels (Other): Group B will be administered insulin at the standard of care levels established by the participating institution.
  Interventions: Other: insulin at the standard of care levels

INTERVENTIONS:
Other: Hyperinsulinemic-normoglycemic clamp — Patients will be randomized to receive the hyperinsulinemic-normoglycemic clamp titrating the blood glucose to 80-110 mg/dL.
  Other Names: clamp; Hyperinsulinemic
  Arms: Hyperinsulinemic-normoglycemic clamp
Other: insulin at the standard of care levels — Subjects will be administered insulin at the standard of care levels established by the participating institution.
  Other Names: insulin
  Arms: Insulin at the standard of care levels

SUMMARY:
Patients undergoing cardiac surgery will be randomized into one of two groups. Group A will be administered insulin using the hyperinsulinemic-normoglycemic clamp to normalize blood glucose levels intra-operatively. Group B will be administered insulin at the standard of care levels established by the participating institution. Patients will be followed at 10 days, 15 days and one year post-operatively.

DETAILED DESCRIPTION:
Using a randomized, controlled design, we propose to test the primary hypothesis that normalization of blood glucose using a hyperinsulinemic-normoglycemic clamp technique reduces the risk of a composite outcome (one or more) of 30-day postoperative mortality and serious postoperative cardiac, renal, neurologic, and infectious postoperative complications in patients undergoing cardiac surgery.

Our secondary hypothesis is that hyperinsulinemic normoglycemic therapy will reduce length of stay in intensive care unit, atrial dysrhythmias, creatinine elevation, hospital readmission, all-cause and cardiac one-year mortality.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-90 years old
* Scheduled for cardiac surgery requiring cardiopulmonary bypass

Exclusion Criteria:

* Off-pump surgical procedures
* Anticipated deep hypothermic circulatory arrest
* In available, baseline cardiac troponin I (>0.5 ng/L) or troponin T (> 0.1 ng/mL) levels (at RVH or CC, respectively)
* Any contraindications to the proposed interventions
* Active infection, including patients with endocarditis or infected pacemaker leads.
* Any infection requiring long- term antibiotics ( > 14 days)
* kidney disease requiring renal replacement therapy

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1439 (Actual)
Dates: Start 2007-07 (Actual); Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andra I Duncan, M.D., Principal Investigator — The Cleveland Clinic; Daniel I Sessler, M.D., Study Director — The Cleveland Clinic; Thomas Schricker, MD, Principal Investigator — Royal Victoria Hospital, Montreal, Canada; George Carvalho, MD, Principal Investigator — Royal Victoria Hospital, Montreal, Canada
Locations (2):
- Cleveland Clinic, Cleveland, Ohio, United States
- Royal Victoria Hospital, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Albacker TB, Carvalho G, Schricker T, Lachapelle K. Myocardial protection during elective coronary artery bypass grafting using high-dose insulin therapy. Ann Thorac Surg. 2007 Dec;84(6):1920-7; discussion 1920-7. doi: 10.1016/j.athoracsur.2007.07.001. PMID 18036907
- [Result] Duncan AE, Kateby Kashy B, Sarwar S, Singh A, Stenina-Adognravi O, Christoffersen S, Alfirevic A, Sale S, Yang D, Thomas JD, Gillinov M, Sessler DI. Hyperinsulinemic Normoglycemia Does Not Meaningfully Improve Myocardial Performance during Cardiac Surgery: A Randomized Trial. Anesthesiology. 2015 Aug;123(2):272-87. doi: 10.1097/ALN.0000000000000723. PMID 26200180
- [Derived] Bellon F, Sola I, Gimenez-Perez G, Hernandez M, Metzendorf MI, Rubinat E, Mauricio D. Perioperative glycaemic control for people with diabetes undergoing surgery. Cochrane Database Syst Rev. 2023 Aug 1;8(8):CD007315. doi: 10.1002/14651858.CD007315.pub3. PMID 37526194
- [Derived] Schricker T, Sato H, Beaudry T, Codere T, Hatzakorzian R, Pruessner JC. Intraoperative maintenance of normoglycemia with insulin and glucose preserves verbal learning after cardiac surgery. PLoS One. 2014 Jun 18;9(6):e99661. doi: 10.1371/journal.pone.0099661. eCollection 2014. PMID 24941010

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Hyperinsulinemic-normoglycemic Clamp | Insulin at the Standard of Care Levels
Started | 709 | 730
Completed | 709 | 730
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Hyperinsulinemic-normoglycemic Clamp | Insulin at the Standard of Care Levels | Total
Number analyzed (Participants) | 709 | 730 | 1439
Age, Continuous [Mean (Standard Deviation); unit: years] | 66 (11) | 66 (11) | 66 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 189 | 184 | 373
  Male | 520 | 546 | 1066
Region of Enrollment [Count of Participants; unit: Participants]
  Canada | 457 | 464 | 921
  United States | 252 | 266 | 518

OUTCOME MEASURES:

1. Primary Outcome: Any Major Morbidity/30-day Mortality
Description: a composite (any versus none) of the following major postoperative complications occurring:
  1. all-cause postoperative mortality
  2. failure to wean from cardiopulmonary bypass or postoperative low cardiac index requiring mechanical circulatory support with intraaortic balloon counterpulsation, ventricular assist device, and/or extracorporeal mechanical oxygenation
  3. serious postoperative infection
  4. acute postoperative kidney injury requiring renal replacement therapy;
  5. new postoperative focal or global neurologic deficit.
Time Frame: within 30 days post surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Hyperinsulinemic-normoglycemic Clamp | Insulin at the Standard of Care Levels
Number analyzed (Participants) | 709 | 730
Participants | 46 | 82
Statistical Analysis 1: Comparison: Hyperinsulinemic-normoglycemic Clamp vs Insulin at the Standard of Care Levels; Test type: Superiority or Other; p = 0.0043, Cochran-Mantel-Haenszel — P-values for combined sites: significant if P < 0.0085 for efficacy. Adjusted for interim analysis. Confidence intervals adjusted for interim analysis; Risk Ratio (RR) = 0.62, 95% CI 2-sided [0.39 to 0.97] — Hyperinsulinemic-normoglycemic clamp

2. Secondary Outcome: Post Operative Atrial Fibrillation
Description: Evidence suggests that maintaining intra-operative normoglycemia during cardiac surgery while providing exogenous glucose and high-dose insulin may decrease post-operative morbidity or mortality. Using a randomized, controlled design, we propose to test the primary hypothesis that normalization of blood glucose using a hyperinsulinemic-normoglycemic clamp technique reduces the risk of a composite of serious adverse outcomes in patients undergoing cardiac surgery
Time Frame: 15 - 30 days post operative
Measure: Count of Participants; unit: Participants
Arm/Group | Hyperinsulinemic-normoglycemic Clamp | Insulin at the Standard of Care Levels
Number analyzed (Participants) | 709 | 730
Participants | 209 | 235
Statistical Analysis 1: Comparison: Hyperinsulinemic-normoglycemic Clamp vs Insulin at the Standard of Care Levels; Test type: Superiority or Other; p = 0.29, Cochran-Mantel-Haenszel; Risk Ratio (RR) = 0.92, 95% CI 2-sided [0.75 to 1.13] — HN vs. standard

3. Secondary Outcome: Duration of Hospitalization
Description: Days from date of surgery to hospital discharge
Time Frame: starting post operative day one to discharge from hospital, on an average of 8 days
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Hyperinsulinemic-normoglycemic Clamp | Insulin at the Standard of Care Levels
Number analyzed (Participants) | 686 | 713
days | 8 [6 to 12] | 8 [6 to 12]
Statistical Analysis 1: Comparison: Hyperinsulinemic-normoglycemic Clamp vs Insulin at the Standard of Care Levels; Test type: Superiority or Other; p = 0.99, Regression, Cox; Hazard Ratio (HR) = 1.05, 95% CI 2-sided [0.91 to 1.21]

4. Secondary Outcome: Duration of Intensive Care Stay
Description: Hours from date of surgery to discharge from intensive care unit
Time Frame: ICU stay hours during hospital stay after surgery, on average of 25 hours
Measure: Median (95% Confidence Interval); unit: hours
Arm/Group | Hyperinsulinemic-normoglycemic Clamp | Insulin at the Standard of Care Levels
Number analyzed (Participants) | 649 | 671
hours | 25 [24.9 to 26.3] | 27 [25.2 to 27.3]
Statistical Analysis 1: Comparison: Hyperinsulinemic-normoglycemic Clamp vs Insulin at the Standard of Care Levels; Test type: Superiority or Other; p = 0.025, Regression, Cox; Risk Ratio (RR) = 1.13, 95% CI 2-sided [0.98 to 1.31] — HN vs. Standard

5. Secondary Outcome: All-cause Mortality
Description: All-cause mortality identified during one-year follow-up.
Time Frame: one year post operative
Measure: Count of Participants; unit: Participants
Arm/Group | Hyperinsulinemic-normoglycemic Clamp | Insulin at the Standard of Care Levels
Number analyzed (Participants) | 653 | 682
Participants | 32 | 22
Statistical Analysis 1: Comparison: Hyperinsulinemic-normoglycemic Clamp vs Insulin at the Standard of Care Levels; Test type: Superiority or Other; p = 0.12, Cochran-Mantel-Haenszel; Risk Ratio (RR) = 1.52, 95% CI 2-sided [0.74 to 3.11] — HN vs. standard

6. Secondary Outcome: a Composite of Minor Postoperative Complications
Description: a composite of minor postoperative complications, which includes: a) prolonged mechanical ventilation, b) low cardiac index, c) acute kidney injury, d) prolonged hospitalization, and 3) all-cause hospital readmission within 30 days.
Time Frame: within 30 days after surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Hyperinsulinemic-normoglycemic Clamp | Insulin at the Standard of Care Levels
Number analyzed (Participants) | 709 | 730
Participants | 200 | 237
Statistical Analysis 1: Comparison: Hyperinsulinemic-normoglycemic Clamp vs Insulin at the Standard of Care Levels; Test type: Superiority or Other; p = 0.085, Cochran-Mantel-Haenszel; Risk Ratio (RR) = 0.88, 95% CI 2-sided [0.72 to 1.07] — HN vs. Standard

ADVERSE EVENTS:
Time Frame: One Year Post-opeperative follow-up for All-Cause Mortality; 1 month Post-opeperative follow-up for Serious Adverse Events and Other (Not Including Serious) Adverse Events
Arm/Group | Hyperinsulinemic-normoglycemic Clamp | Insulin at the Standard of Care Levels
All-Cause Mortality (participants affected / at risk) | 32/709 | 22/730
Serious Adverse Events (participants affected / at risk) | 18/709 | 27/730
Other Adverse Events (participants affected / at risk) | 0/709 | 0/730
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Hyperinsulinemic-normoglycemic Clamp (N=709) | Insulin at the Standard of Care Levels (N=730)
sae (Surgical and medical procedures) | 18 (18) | 27 (27) — Adverse Events were monitored/assessed without regard to the specific Adverse Event Term

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No